CLINICAL TRIAL: NCT03238703
Title: An Investigator Initiated Registry of Simple Oral Therapy for Low Risk Breast Cancer (SOLR)
Brief Title: Endocrine Therapy in Treating Patients With HER2 Negative, Low Risk Breast Cancer
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Administrative closure based on sponsor recommendation, prior to subject enrollment
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9764; NCI-2017-00724 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9764 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2017-07-31; First posted 2017-08-03 (Actual); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: HER2/Neu Negative; Invasive Breast Carcinoma; Postmenopausal; Stage 0 Breast Cancer; Stage IA Breast Cancer
MeSH Terms: conditions — Breast Carcinoma In Situ; Breast Neoplasms | interventions — Anastrozole; exemestane; Letrozole; Tamoxifen; Toremifene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (AI, SERM) (Experimental): Patients receive exemestane PO QD, anastrozole PO QD, letrozole PO QD, tamoxifen citrate PO QD, or toremifene citrate PO QD at the discretion of the treating physician. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Anastrozole; Drug: Exemestane; Other: Laboratory Biomarker Analysis; Drug: Letrozole; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Tamoxifen Citrate; Drug: Toremifene Citrate

INTERVENTIONS:
Drug: Anastrozole — Given PO
  Other Names: Anastrazole; Arimidex; ICI D1033; ICI-D1033; ZD-1033
Drug: Exemestane — Given PO
  Other Names: Aromasin; FCE-24304
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Letrozole — Given PO
  Other Names: CGS 20267; Femara
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Drug: Tamoxifen Citrate — Given PO
  Other Names: Apo-Tamox; Clonoxifen; Dignotamoxi; Ebefen; Emblon; Estroxyn; Fentamox; Gen-Tamoxifen; Genox; ICI 46,474; ICI-46474; Jenoxifen; Kessar; Ledertam; Lesporene; Nolgen; Noltam; Nolvadex; Nolvadex-D; Nourytam; Novo-Tamoxifen; Novofen; Noxitem; Oestrifen; Oncotam; PMS-Tamoxifen; Soltamox; TAM; Tamax; Tamaxin; Tamifen; Tamizam; Tamofen; Tamoxasta; Tamoxifeni Citras; Zemide
Drug: Toremifene Citrate — Given PO
  Other Names: Acapodene; Fareston; FC-1157a; GTx-006

SUMMARY:
This pilot clinical trial studies how well endocrine therapy works in treating patients with HER2 negative, low risk breast cancer. Estrogen can cause the growth of breast cancer cells. Endocrine therapies such as aromatase inhibitors and selective estrogen receptor modulators may lessen the amount of estrogen made by the body.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the conversion rate from a standard low-toxicity approach to guideline-directed therapy which includes surgery +/- radiation therapy as a result of progression of disease or patient/provider choice.

II. To examine factors that might differ between those who convert from the low-toxicity approach to the guideline-directed therapy and those do not convert.

SECONDARY OBJECTIVES:

I. To measure the safety and clinical effectiveness of systemic endocrine therapy used in a prolonged neoadjuvant fashion.

II. To evaluate the impact of risk-stratified care in Quality-Adjusted Life Years (QALY) and QALY gains.

III. To estimate the cost savings of indefinitely delaying surgery and radiation in favor of systemic endocrine therapy alone.

OUTLINE:

Patients receive exemestane orally (PO) once daily (QD), anastrozole PO QD, letrozole PO QD, tamoxifen citrate PO QD, or toremifene citrate PO QD at the discretion of the treating physician. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent
* A diagnosis of invasive breast cancer, with or without an in situ component, that is:

  * Originally identified by screening mammography
  * Characterized by standard diagnostic mammography +/- breast ultrasound
  * Clinically node negative
  * Confirmed by breast magnetic resonance imaging (MRI) in a facility that maintains active American College of Radiology (ACR) accreditation to be of low clinical stage (=< 2 cm, node negative, unifocal invasive)
  * Estrogen receptor (ER) and progesterone receptor (PR) Allred scored, each > 5/8
  * Her2 negative using American Society of Clinical Oncology (ASCO)-College of American Pathologists (CAP) guidelines
  * ki-67 proliferation scored, < 20%
  * Clinical Nottingham grade 1 or 2
  * Scored on the MammaPrint 70-gene breast cancer recurrence assay as low risk
* Prior to the discovery of the breast cancer, clinically post-menopausal as defined as: i) one or more years from last menses; or ii) history of oophorectomy; or iii) follicle stimulating hormone (FSH) test result in the post-menopause reference range
* Willing to accept oral endocrine therapy with a third generation aromatase inhibitor (AI) or selective estrogen receptor modifier (SERM)
* Willing to undergo routine surveillance with breast ultrasound and/or mammography

Exclusion Criteria:

* Known contraindication to aromatase inhibitor or SERM therapy
* Pregnant at time of or within prior year of diagnosis
* Clinically detected or palpable disease prior to biopsy in either breast or ipsilateral axilla
* Prior history of invasive breast cancer or ductal breast carcinoma in situ (DCIS)
* Prior use of aromatase inhibitor therapy apart from assisted reproduction
* Prior use of SERM
* Unmanaged/uncontrolled mental health disorder
* Life expectancy < 6 months (m) for any cause
* Biopsy confirmed multifocal, multicentric, or contralateral disease that is invasive or non-invasive
* DCIS with focal invasion

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2023-03-14 (Estimated); Study Completion 2025-03-14 (Estimated)

PRIMARY OUTCOMES:
Conversion from oral endocrine therapy for any reason to guideline-directed therapy | Up to 5 years
  Includes clinical or radiographic progression, patient preference, endocrine therapy intolerance or toxicity, or death from any cause. Descriptive statistics will be summarized among all patients and patients within each of the two groups (stay with oral therapy vs conversion due to any causes).

SECONDARY OUTCOMES:
Advanced imaging (if performed on any subset of patients) | Up to 5 years
  Will be compared to a concurrent group of patients managed in the conventional manner with upfront surgery +/- radiation therapy followed by systemic endocrine therapy. Descriptive statistics will be summarized among all patients and patients within each of the two groups (stay with oral therapy vs conversion due to any causes).
Cost-effectiveness and patient-centeredness outcomes defined as financial toxicity and solubility, quality of life (physical, mental, emotional changes) on endocrine therapy, and, access to support services | Up to 5 years
  Comparisons will be made to historical benchmarks for similar patients managed in a conventional locoregional manner for early-stage breast cancer. Descriptive statistics will be summarized among all patients and patients within each of the two groups (stay with oral therapy vs conversion due to any causes).
Effect of age | Up to 5 years
  Will be compared to a concurrent group of patients managed in the conventional manner with upfront surgery +/- radiation therapy followed by systemic endocrine therapy. Descriptive statistics will be summarized among all patients and patients within each of the two groups (stay with oral therapy vs conversion due to any causes).
Effect of comorbidity severity interaction | Up to 5 years
  Will be compared to a concurrent group of patients managed in the conventional manner with upfront surgery +/- radiation therapy followed by systemic endocrine therapy. Descriptive statistics will be summarized among all patients and patients within each of the two groups (stay with oral therapy vs conversion due to any causes).
Effect of type of endocrine therapy type (selective estrogen receptor modifier versus aromatase inhibitor) | Up to 5 years
  Will be compared to a concurrent group of patients managed in the conventional manner with upfront surgery +/- radiation therapy followed by systemic endocrine therapy. Descriptive statistics will be summarized among all patients and patients within each of the two groups (stay with oral therapy vs conversion due to any causes).
Effects emanating from tertiary care | Up to 5 years
  Will be compared to a concurrent group of patients managed in the conventional manner with upfront surgery +/- radiation therapy followed by systemic endocrine therapy. Descriptive statistics will be summarized among all patients and patients within each of the two groups (stay with oral therapy vs conversion due to any causes).
Progression of disease while on primary endocrine therapy, as measured objectively by routine diagnostic breast imaging (mammography and/or ultrasound) | Up to 5 years
  Descriptive statistics will be summarized among all patients and patients within each of the two groups (stay with oral therapy vs conversion due to any causes).

CONTACTS AND LOCATIONS:
Overall Officials: Vijayakrishna Gadi, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No